CLINICAL TRIAL: NCT06856512
Title: Intradialytic Exercise and Remote Ischaemic Preconditioning: a Cardioprotective Role ?
Acronym: EXPI-DIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Avignon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AU-092024-CM; LAPEC/2024/DIAL (Other: Avignon University)
Record Dates: First submitted 2025-02-05; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; myocardial function; exercise; remote ischemic preconditioning; myocardial stunning; cardioprotection
MeSH Terms: conditions — Motor Activity; Myocardial Stunning | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All patients are randomly assigned to standard dialysis, dialysis with intermittent intradialytic exercise and dialysis with intermittent remote ischaemic preconditioning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients issued from dialysis units (clinic) (Experimental): Randomised, controlled, crossover, bicentric, single-blind, prospective, open-label, superiority clinical trial comparing 3 dialysis modalities:
  Procedure A: Standard dialysis
  Procedure B: Dialysis with intradialytic intermittent physical exercise
  Procedure C: Dialysis with intradialytic ischaemia/reperfusion sequence of the upper limb
  Each subject will realize the 3 sessions in a random order.
  Interventions: Other: Remote ischaemic preconditioning; Other: Exercise; Other: standard dialysis

INTERVENTIONS:
Other: Remote ischaemic preconditioning — The dialysis protocol integrates a sequence of five ischaemia/reperfusion blocks applied to the upper limb. Each block consists of a 5-minute period of cuff inflation at a supra-systolic pressure individualized to each patient-20 mmHg above the limb occlusion pressure-followed by a 25-minute period of cuff deflation. This intervention begins 30 minutes after the start of dialysis and is referred to as hemodialysis remote ischaemic preconditioning (HD-rIPC).
Other: Exercise — The exercise protocol consists of five sequential bouts of physical activity, initiated 30 minutes after the start of dialysis. Each bout comprises a 5-minute cycling exercise at moderate intensity, corresponding to a Borg Scale rating of 12-14, followed by a 25-minute passive recovery phase. This structured intervention is referred to as hemodialysis exercise (HD-EX).
Other: standard dialysis — The hemodialysis control condition (HD-CONT) consists of standard hemodialysis treatment without the integration of any additional interventions, such as exercise or ischaemia/reperfusion protocols.

SUMMARY:
The aim of this clinical trial is to evaluate whether intermittent exercise and remote ischaemic preconditioning (rIPC) during haemodialysis (HD) can provide cardioprotection in adult patients (aged 20-79 years) undergoing HD for at least 3 months. The main questions to be answered are

Does intermittent exercise or rIPC reduce myocardial stunning during HD? Do these interventions have a beneficial effect on haemorheology, arrhythmias, systemic inflammation and HD efficiency? The investigators will compare three HD sessions: no intervention (HD-CONT), with moderate-intensity intermittent exercise (HD-EX), and with rIPC using cuff inflation (HD-rIPC) to see if HD6EX and HD-rIPC approaches offer enhanced cardioprotection.

Participants will:

Undergo three randomised HD sessions. Participate in 5 blocks of moderate-intensity exercise or rIPC during the HD sessions.

Have cardiac function and biomarkers assessed before, during and after HD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 79 years.
* Patients on hemodialysis for more than 3 months.
* No engagement in regular exercise outside of dialysis.
* No prior exposure to intradialytic exercise within the past six months.
* No medical contraindications to physical activity.
* Life expectancy greater than 6 months.
* Patients with relative good echogenicity

Exclusion Criteria

* Patient is participating in another Category I interventional study, or has participated in another interventional study within the past 3 months
* The patient is in an exclusion period determined by a previous study
* The patient is under legal protection or under guardianship or curatorship It turns out to be impossible to give the patient informed information, or the patient refuses to sign the consent
* Pregnant, parturient or breastfeeding patient
* Patients with unstable coronary artery disease.
* Patients with peripheral artery disease (stage III or IV) in the lower limbs.
* Patients with limb amputation.
* Patients with musculoskeletal disorders impairing exercise.
* Presence of a pacemaker, cardiac stimulation device, or implantable cardioverter defibrillator (ICD).
* History of heart transplant.
* Patients with uncontrolled hypertension.
* Refractory anemia.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in regional myocardial stunning. | From enrollment to the end of treatment at 7 weeks
  The investigators will use echocardiography to assess the number of left ventricular myocardial segments (using a 18-segment model), that demonstrate a reduction in longitudinal deformation greater than 20% at peak stress during hemodialysis, relative to baseline measurements obtained at the start of the dialysis session. Their aim is to compare changes in regional wall motion abnormalities across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.

SECONDARY OUTCOMES:
Hemorheology - blood viscosity | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in whole blood viscosity, measured using a cone-plate viscometer, from the beginning to the peak stress of dialysis. Their aim is to compare these changes in whole blood viscosity across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of dialysis and just before its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Hemorheology - erythrocyte deformability | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in erythrocyte deformability, measured using an ektacytometer, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of dialysis and just before its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Hemorheology - erythrocyte aggregation | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in erythrocyte aggregation, measured using an ektacytometer, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of dialysis and just before its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - fibrinogen | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in fibrinogen, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of dialysis and just before its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - miRNA | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in levels of circulating mi-RNAs, quantified by reverse transcription-quantitative polymerase chain reaction (RT-qPCR), from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Intraventricular pressure gradient | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in the left intraventricular pressure gradient, measured by postprocessing color Doppler M-mode echocardiographic images, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Hemodynamic parameters - cardiac output | From enrollment to the end of treatment at 7 weeks
  The investigators will measure cardiac output every 30minutes from the beginning to the end of dialysis during the 3 conditions. Their aim is to compare the changes during HD across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). For HD-EX and HD-RIPC, the investigators will add a measure immediately after the interventions (exercise or vascular occlusion) to control for the effect of the intervention. Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Hemodynamic parameters - blood pressure | From enrollment to the end of treatment at 7 weeks
  The investigators will measure blood pressure every 30minutes from the beginning to the end of dialysis during the 3 conditions. Their aim is to compare the changes during HD across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). For HD-EX and HD-RIPC, the investigators will add a measure immediately after the interventions (exercise or vascular occlusion) to control for the effect of the intervention. Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Intraventricular flow | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in the velocity vector fields of blood flow in the LV, calculated by postprocessing color Doppler echocardiographic images, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Sublingual microvasculature - proportion of perfused vessels | From enrollment to the end of treatment at 7 weeks
  The investigators will assess the variation in the proportion of perfused vessels, measured using a videomicroscope, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Sublingual microvasculature - functional capillary density | From enrollment to the end of treatment at 7 weeks
  The investigators will assess the variation in functional capillary density, measured using a videomicroscope, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Sublingual microvasculature - De Baker's score | From enrollment to the end of treatment at 7 weeks
  The investigators will assess the variation in De Baker's score, measured using a videomicroscope, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Sublingual microvasculature - per-capillary microcirculatory flow index | From enrollment to the end of treatment at 7 weeks
  The investigators will assess the variation in per-capillary microcirculatory flow index, measured using a videomicroscope, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Sublingual microvasculature - red blood cell mean velocity | From enrollment to the end of treatment at 7 weeks
  The investigators will assess the variation in red blood cell mean velocity, measured using a videomicroscope, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Sublingual microvasculature - total vessel density | From enrollment to the end of treatment at 7 weeks
  The investigators will assess the variation in total vessel density, measured using a videomicroscope, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
standard echocardiography - LA morphology and function | From enrollment
  The investigators will evaluate the left atrial (LA) volumes during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the LA morphology and function of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - LV volumes | From enrollment
  The investigators will evaluate the left ventricular (LV) volumes using echocardiography during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - LV global diastolic function - E wave | From enrollment to the end of treatment at 7 weeks
  The investigators will evaluate the variation in E wave by pulsed Doppler ehocardiography from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
standard echocardiography - LV global diastolic function - tricuspid regurgitation | From enrollment
  The investigators will evaluate the tricuspid regurgitation by continuous-wave Doppler ehocardiography during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. It will be used to characterize left ventricular global diastolic function. Measurements will be conducted 30 minutes before the onset of dialysis
standard echocardiography - RV systolic function - TAPSE | From enrollment
  The investigators will evaluate the Tricuspid Annular Plane Systolic Excursion using echocardiography during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. It will be used to characterize right ventricular global systolic function. Measurements will be conducted 30 minutes before the onset of dialysis
standard echocardiography - RV morphology - areas | From enrollment
  The investigators will evaluate the right ventricular (RV) area at end-systole and end-diastole during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - RV global diastolic function - Et wave | From enrollment
  The investigators will evaluate the Et wave by pulsed Doppler ehocardiography during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. It will be used to characterize right ventricular global diastolic function. Measurements will be conducted 30 minutes before the onset of dialysis
Biological data - uraemic toxins - beta2-microglobulin | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in beta2-microglobulin level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - uraemic toxins - Indoxyl sulfate | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in indoxyl sulfate level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - uraemic toxins - p-Cresyl sulfate | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in p-Cresyl sulfate level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - uraemic toxins - myoglobin | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in myoglobin level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - uraemic toxins - free light chains | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in free light chains, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - cardiac biomarkers - NT-pro-BNP | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in NT-pro-BNP level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - cardiac biomarkers - BNP level | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in BNP level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - cardiac biomarkers - cardiac troponin T | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in cardiac troponin T level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - cardiac biomarkers - sST2 | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in levels of soluble ST2, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
biological data - characterization of patients - sodium | From enrollment
  The investigators will evaluate the blood level of sodium during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - potassium | From enrollment
  The investigators will evaluate the serum level of potassium during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - calcium | From enrollment
  The investigators will evaluate the serum level of calcium during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - phosphate | From enrollment
  The investigators will evaluate the serum level of phosphate during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - vitamin D | From enrollment
  The investigators will evaluate the serum level of vitamin D during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - parathyroid hormone | From enrollment
  The investigators will evaluate the serum level of parathyroid hormone during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - creatinine | From enrollment
  The investigators will evaluate the serum level of creatinine during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - creatinine clearance | From enrollment
  The investigators will evaluate the creatinine clearance during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - urea | From enrollment
  The investigators will evaluate the blood level of urea during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - Kt/V | From enrollment
  The investigators will evaluate the Kt/V urea during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients.
biological data - characterization of patients - nPCR | From enrollment
  The investigators will evaluate the normalized proteïn catabolic rate during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - albumin | From enrollment
  The investigators will evaluate the serum level of albumin during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - characterization of patients - CRP | From enrollment
  The investigators will evaluate the serum level of c-reactiv protein during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the progression of the disease in the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - hematology - complete blood count | From enrollment
  The investigators will evaluate the complete blood count during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the blood of patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - hematology - ferritin | From enrollment
  The investigators will evaluate the serum ferritin level during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the blood of patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - hematology - transferrin saturation | From enrollment
  The investigators will evaluate the transferrine saturation during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the blood of patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Hematology - hematocrit | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in hematocrit, measured using an hemoglobinometer, from the beginning to the peak stress of dialysis. Their aim is to compare these changes in whole blood viscosity across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Hematology - hemoglobin | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in hemoglobin level, measured using an hemoglobinometer, from the beginning to the peak stress of dialysis. Their aim is to compare these changes in whole blood viscosity across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
biological data - lipidic profile - LDL cholesterol | From enrollment
  The investigators will evaluate the LDL cholesterol during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the lipidic profile. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - lipidic profile - HDL cholesterol | From enrollment
  The investigators will evaluate the HDL cholesterol during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the lipidic profile of patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - lipidic profile - triglycerides | From enrollment
  The investigators will evaluate the triglycerides level during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrolment. They will be used to characterize the lipidic profile of patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Biological data - inflamation - ultra-sensitive c-reactive protein | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in ultra-sensitive c-reactive protein level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of the dialysis and at its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - inflamation - interleukin-6 | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in interleukin-6 level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of the dialysis and at its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - inflamation - interleukin-10 | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in interleukin-10 level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of the dialysis and at its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - inflamation - tumor necrosis factor-α | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in tumor necrosis factor-α level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of the dialysis and at its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - endothelial cell activation - intercellular adhesion molecule-1 | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in intercellular adhesion molecule-1 level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of the dialysis and at its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - endothelial cell activation - vascular cell adhesion molecule-1 | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in vascular cell adhesion molecule-1 level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of the dialysis and at its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - endothelial cell activation - endothelin | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in endothelin level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of the dialysis and at its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Biological data - endothelial cell activation - proendothelin | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in proendothelin level, measured by analysing blood sample, from the beginning to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset of the dialysis and at its end. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
biological data - insulin resistance - glucose | From enrollment
  The investigators will evaluate the glucose level during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to quantify the insulin resistance of patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - insulin resistance - glycated hemoglobin | From enrollment
  The investigators will evaluate the glycated hemoglobin level during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to quantify the insulin resistance of patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
biological data - insulin resistance - insulin | From enrollment
  The investigators will evaluate the insulin level during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to quantify the insulin resistance of patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Hemodynamic parameters - heart rate | From enrollment to the end of treatment at 7 weeks
  The investigators will measure heart rate every 30minutes from the beginning to the end of dialysis during the 3 conditions. Their aim is to compare the changes during HD across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). For HD-EX and HD-RIPC, the investigators will add a measure immediately after the interventions (exercise or vascular occlusion) to control for the effect of the intervention. Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Hemodynamic parameters - stroke volume | From enrollment to the end of treatment at 7 weeks
  The investigators will measure stroke volume every 30minutes from the beginning to the end of dialysis during the 3 conditions. Their aim is to compare the changes during HD across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). For HD-EX and HD-RIPC, the investigators will add a measure immediately after the interventions (exercise or vascular occlusion) to control for the effect of the intervention. Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Strains - LV | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in left longitudinal strains, using speckle tracking echocardiography, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Strains (in %) measure the amount of myocardial longitudinal shortening of the cavity, are relatively load-independent, and can detect subclinical myocardial dysfunction, even when it is not apparent by conventional echocardiography.
  Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Strains - RV | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in right ventricular longitudinal strains, using speckle tracking echocardiography, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Strains (in %) measure the amount of myocardial longitudinal shortening of the cavity, are relatively load-independent, and can detect subclinical myocardial dysfunction, even when it is not apparent by conventional echocardiography.
  Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Strains - LA | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in left atrial longitudinal strains, using speckle tracking echocardiography, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Strains (in %) measure the amount of myocardial longitudinal shortening of the cavity, are relatively load-independent, and can detect subclinical myocardial dysfunction, even when it is not apparent by conventional echocardiography.
  Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
standard echocardiography - LV morphology - diameter | From enrollment
  The investigators will evaluate the left ventricular (LV) diameter at both end-diastole and end-systole during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the LV morphology of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - LV morphology - wal thicknessess | From enrollment
  The investigators will evaluate the left ventricular (LV) wall thicknesses at both end-diastole and end-systole during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the LV morphology of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - RV morphology - diameters | From enrollment
  The investigators will evaluate the right ventricular (RV) diameters at end-systole and end-diastole during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the RV morphology of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - LV global systolic function | From enrollment
  The investigators will evaluate the left ventricular (LV) ejection fraction using echocardiography during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to evaluate the LV global systolic function. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - LV morphology - mass | From enrollment
  The investigators will evaluate the left ventricular (LV) mass during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the LV morphology of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
Myocardial work - global myocardial work | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in global myocardial work, using speckle tracking echocardiography and blood pressure, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). It provides a more precise assessment of cardiac performance than strains by considering the left ventricular loading condition. Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Myocardial work - global constructive work | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in global constructive work, using speckle tracking echocardiography and blood pressure, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). It provides a more precise assessment of cardiac performance than strains by considering the left ventricular loading condition. Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Myocardial work - global wasted work | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in global wasted work, using speckle tracking echocardiography and blood pressure, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). It provides a more precise assessment of cardiac performance than strains by considering the left ventricular loading condition. Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
Myocardial work - global work efficiency | From enrollment to the end of treatment at 7 weeks
  The investigators will assess variations in global work efficiency, using speckle tracking echocardiography and blood pressure, from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). It provides a more precise assessment of cardiac performance than strains by considering the left ventricular loading condition. Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
standard echocardiography - LV global diastolic function - A wave | From enrollment to the end of treatment at 7 weeks
  The investigators will evaluate the variation in A wave measured by pulsed Doppler ehocardiography from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
standard echocardiography - RV systolic function | From enrollment
  The investigators will calculate the right ventricular fractional area change using echocardiography during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. It will be used to characterize right ventricular global systolic function. Measurements will be conducted 30 minutes before the onset of dialysis
standard echocardiography - RV global diastolic function | From enrollment
  The investigators will evaluate the At wave by pulsed Doppler ehocardiography during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. It will be used to characterize right ventricular global diastolic function. Measurements will be conducted 30 minutes before the onset of dialysis
standard echocardiography - tissue Doppler imaging - LV e' | From enrollment
  The investigators will evaluate the left ventricular (LV) e' wave by tissue Doppler imaging during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the LV regional function of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - tissue Doppler imaging - LV a' | From enrollment
  The investigators will evaluate the left ventricular (LV) a' wave by tissue Doppler imaging during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the LV function of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - tissue Doppler imaging - LV s' | From enrollment
  The investigators will evaluate the left ventricular (LV) s' waves by tissue Doppler imaging during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the LV regional function of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - tissue Doppler imaging - RV e' | From enrollment
  The investigators will evaluate the right ventricular (RV) e' wave by tissue Doppler imaging during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the RV regional function of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - tissue Doppler imaging- RV a' | From enrollment
  The investigators will evaluate the right ventricular (RV) a' wave by tissue Doppler imaging during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the RV regional function of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - tissue Doppler imaging - RV s' | From enrollment
  The investigators will evaluate the right ventricular (RV) s' wave by tissue Doppler imaging during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the RV regional function of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - RV morphology and function - diameters | From enrollment
  The investigators will evaluate the right ventricular (RV) outflow tract diameters during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the RV morphology and function of the patients. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - RV global diastolic function - Et/At ratio | From enrollment
  The investigators will evaluate the Et/At ratio by pulsed Doppler ehocardiography during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. It will be used to characterize right ventricular global diastolic function. Measurements will be conducted 30 minutes before the onset of dialysis
standard echocardiography - LV global diastolic function - E/A | From enrollment to the end of treatment at 7 weeks
  The investigators will evaluate the E/A ratio by pulsed Doppler ehocardiography from before to the peak stress of dialysis. Their aim is to compare these changes across three experimental conditions: - Standard hemodialysis (HD-CONT), - Hemodialysis with intradialytic intermittent physical exercise (HD-EX), - Hemodialysis with an intradialytic ischemia/reperfusion sequence applied to the upper limb (HD-RIPC). Patients will participate in all three conditions in a randomized order. A two-week period of standard dialysis will separate the execution of two consecutive sessions.
standard echocardiography - diastolic function - LV E/e' | From enrollment
  The investigators will evaluate the left ventricular (LV) E/e' ratio during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the LV filling pressure. Measurements will be conducted 30 minutes before the onset of dialysis.
standard echocardiography - diastolic function - RV Et/e' | From enrollment
  The investigators will evaluate the right ventricular (RV) Et/e' ratio during the first dialysis session (HD-CONT, HD-EX, or HD-rIPC, depending on the randomized order of the three sessions), after enrollment. They will be used to characterize the RV filling pressure. Measurements will be conducted 30 minutes before the onset of dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Laure Patrier, MD, PhD, Principal Investigator — AIDER Santé - Fondation Charles Mion
Locations (3):
- France (3):
  - Aider Sante, Montpellier
  - Aider Sante, Nîmes
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No